CLINICAL TRIAL: NCT03365505
Title: Frailty Assessment in Elderly Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00-34-17-MMC
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Frail Elderly Syndrome; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is known as an independent risk factor for morbidity and mortality in older cardiac patients . It is an important factor on the cardiologist decision between conservative and invasive treatment in older patient with acute coronary syndrome, and is usually made subjectively by the cardiologist known in the literature as eyeball testing.

in this study the investigators will compare the cardiologists eye ball testing to objective frailty assessment based on Fried score and Edmonton frailty scale.

DETAILED DESCRIPTION:
elderly patients admitted to Meir hospital with acute coronary syndrome will be assessed for frailty twice: the first frailty assessment will be a subjective eye ball testing made by the cardiologist, the second assessment will be an objective one based on Fried frailty score and Edmonton frail scale.

The cardiologist will not be aware of the objective frailty assessment result.

The eye ball testing will be compared to the objective frailty assessment (Fried score and Edmonton frailty scale).

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to Meir hospital with acute coronary syndrome
* Age: 80 years old and older
* eligible for signing an informed concent

Exclusion Criteria:

* uncontrolled heart failure ( pulmonary edema or the use of iv diuretics)
* cardiogenic shock
* fever st elevation myocardial infarction

Ages: 80 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patient admitted to our hospital with acute coronary syndrome: unstable angina or non ST elevation myocardial infarction who are aged 80 and above and are hemodinamically stable.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
A subjective eye ball frailty assessment will be compared to an objective frailty assessment based on Fried score and Edmonton frailty scale | Through hospitalization , an average of 1 week
  Subjective frailty assessment made by a cardiologist during hospitalization with acute coronary syndrome- "eye ball" testing
An objective frailty assessment using Fried score and Edmonton frailty scale will be compared to a subjective eye ball frailty assessment | Through hospitalization , an average of 1 week
  An objective frailty assessment based on Fried score and Edmonton frailty scale